CLINICAL TRIAL: NCT05088993
Title: Effects of Antigravity Treadmill Training on Gait and Balance in Patients With Diabetic Polyneuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Shamekh Mohamed El-Shamy, Professor, Umm Al-Qura University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Umm AlQura Un.
Record Dates: First submitted 2021-10-07; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Diabetic Polyneuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antigravity Treadmill Group (Experimental): This group received antigravity treadmill training 100% weight bearing and conventional exercise program.
  Interventions: Other: Antigravity treadmill training; Other: Conventional exercise program
- Conventional Exercise Group (Active Comparator): This group received the conventional exercise program only.
  Interventions: Other: Conventional exercise program

INTERVENTIONS:
Other: Antigravity treadmill training — This group received antigravity treadmill training 100% weight bearing
  Arms: Antigravity Treadmill Group
Other: Conventional exercise program — This group received the conventional exercise program only.

SUMMARY:
Aging can be defined as sequential deterioration that occurs in elderly people including weakness, loss of mobility, decline of physical capabilities, increase susceptibility to disease and many other age-related physiological changes .The beginning of old age in most developed countries is about 60 or 65 years old. Diabetes mellitus (DM) and most commonly type 2 DM is one of the most common chronic non-communicable diseases affecting old people in Saudi Arabia which might be resulted from decline in physical activities. Polyneuropathy (PN) and its serious consequences represent the most common complication in diabetic mellitus which could contribute to an increased gait abnormality and risk of falling.

DETAILED DESCRIPTION:
Disability and reduction of quality of life are the largest costs of diabetes and its complications. So taking active intervention to reduce the risk of falls, improve gait performance and improve the quality of life in elderly with DPN is very important. Lower extremity aerobic exercise training via treadmill aiming for improving patients' physical activity levels is an important part in the rehabilitation program to enhance balance and walking functions and reducing the fall risk, .Treadmill training using s low-load walking provided by an emerging technology called lower body positive pressure (LBPP) that effectively reduces body weight could be preferable than other methods of unweighting treadmill because the air pressure is applied uniformly over the lower body. This kind of anti-gravity treadmill is ideal in reducing the formation of pain and pressure points that are common with harness-based unweighting systems. Many other advantages are also associated with this unique type of antigravity technology that could give it the superiority than the other types of unweighting treadmills in enhancing walking performance, reducing the risk of fall and improving quality of life in Saudi elderly people with DPN.

ELIGIBILITY:
Inclusion Criteria:

* Elderly Saudi men with diabetic polyneuropathy with history of 2 or more falls within the past 12 months
* Diagnosed as having uncontrolled Type 2 Diabetes Mellitus, with glycosylated hemoglobin (HbA1c) level between 7 and 11 and fasting glucose level ranged from 7.0 -11.1 mmol/L.
* Treated only with oral anti-diabetic agents (not taking insulin),
* Pharmacological treatment had to be stable for at least 3 months before the study.
* They will be selected among old subjects that were able to walk independently with or without assistive device, but with poor balance

Exclusion Criteria:

* Type 1 Diabetes Mellitus,
* Patients who had got a score over 19 according to Tinetti scale of balance assessment,
* Patient with malnutrition (BMI < 21 kg/m2 or with recent weight loss > 5% body weight in the last month or > 10% in six months),
* Patients with established hypertension (resting systolic blood pressure > 140 mm Hg and diastolic blood pressure > 90 mm Hg,
* With any severe chronic or uncontrolled comorbid condition as recent myocardial infarction, unstable angina, acute congestive heart failure, third degree heart block and uncontrolled arrhythmia.
* Patients will be excluded also if they have abnormal skin integrity e.g. wound or scar tissues or are on other complementary treatment,
* History of serious cerebrovascular or cardiovascular diseases, and severe debilitating musculoskeletal problems).

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline spatial and temporal gait parameters at 3 months | Baseline and 3 months post-intervention
  Spatial and temporal gait analysis will be evaluated for every patient at baseline and 3 months post-intervention by using the 3-D motion analysis system.
Change from baseline postural stability at 3 months | Baseline and 3 months post-intervention
  Postural stability assessment by using Balance Biodex stability system measuring (antero-posterior, medio-lateral, and overall stability indices.

SECONDARY OUTCOMES:
Change from baseline functional capacity at 3 months | Baseline and 3 months post-intervention
  The assessment of functional capacity will be done using Six Minute Walk Test where intensity is moderately higher than daily living activities. Subject will be asked to walk at his own maximal pace from end to end of a 40-meter flat, straight corridor marked every 1 meter with side cones, in order to cover as much ground as possible while maintaining a steady pace without running during the allowed time. No verbal encouragement will be given, and subjects will be informed verbally each 2 minutes of the remaining time. The patients will be allowed to stop, but they can start again, if possible, within the allocated 6 minutes. Distance covered in 6 minutes will be recorded in meter. The longer the distance that will be walked will signify a better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Shamekh M Elshamy, Ph.D., Principal Investigator — Professor
Locations (1):
- Al Noor Specialized Hospital, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No